CLINICAL TRIAL: NCT04218825
Title: Study to Determine the Aetiology of Chlormethine Gel Induced-skin Drug Reaction in Early Stage Mycosis Fungoides Cutaneous T Cell Lymphoma (MF-CTCL)
Brief Title: REACH: Study to Determine the Aetiology of Chlormethine Gel Induced-skin Drug Reaction in Early Stage Mycosis Fungoides Cutaneous T Cell Lymphoma (MF-CTCL)
Acronym: REACH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After an extensive assessment of the study feasibility, it was decided to discontinue the clinical trial due to poor recruitment.
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1754-CLTF; 2019-004891-20 (EudraCT Number)
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-09

CONDITIONS: Early Stage Mycosis Fungoides Cutaneous T Cell Lymphoma (MF-CTCL) (Stage IA-IB)
Keywords: mycosis fungoides (MF); cutaneous T cell lymphoma (CTCL)
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with early stage MF-CTCL (stage IA-IB) (Experimental): Patients are treated with Chlormethine gel (CL) gel. In case of any skin drug reaction, allergic test will be carried out. Patients not allergic to CL gel will continue at reduced application frequency, with the addition of topical steroid if necessary.
  Interventions: Drug: chlormethine gel

INTERVENTIONS:
Drug: chlormethine gel — Gel to be applied to all skin areas affected by MF-CTCL
  Other Names: Ledaga®

SUMMARY:
Adult patients with early stage MF-CTCL (stage IA-IB) will be eligible for this study. A total of 100 early stage MF-CTCL patients diagnosed in the past year will be enrolled.

Treatment with CL gel will be applied once daily to all skin areas affected by MF-CTCL and, for 8 weeks, one selected skin area unaffected by MF-CTCL (0.5% body surface area) until treatment response (complete response), study treatment duration completed (56 weeks), progression, or another withdrawal criterion is met.

Depending on the type of skin drug-related reaction (if any) occurring after application of CL gel, this study will categorize patients into three different groups corresponding to three different treatment patterns:

* Group A: Patients with no skin drug reaction with CL gel application
* Group B: Patients developing a skin drug reaction of any grade with CL gel application, not due to allergic reaction to CL gel, will continue treatment at reduced application frequency
* Group C: Patients from Group B unable to tolerate reduced CL gel application frequency will apply a potent topical steroid twice daily in addition to CL gel applied every other day

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MF-CTCL stage IA or IB at enrolment as per ISCL/EORTC revision to the MF and Sézary syndrome classification and MF stage should have never met the criteria for stage IIA or higher in the patient medical history
* Lesions cover less than 80% of BSA
* Age ≥ 18
* ECOG/WHO performance status 0-2

Exclusion Criteria:

* Previous treatment with CL gel
* Concurrent or planned local or systemic anti-CTCL therapy
* Prior treatment with antihistamines or narrow band UV-B or PUVA therapy one week before enrolment, or systemic corticosteroids or radiotherapy in the last 4 weeks before enrolment
* Prior treatment with topical steroids in the patch test area (upper back) one week before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) for all patients and in groups A, B and C. | 2.5 years from first patient in
  The response status - complete response (CR), partial response (PR), stable disease (SD) and disease progression (PD) - will be assessed using the global response assessment: skin, lymph nodes (not involved at entry), viscera (not involved at entry) and blood (absolute value CD4+CD7- and CD4+CD26- circulating population) as per EORTC-ISCL-USCLC guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Julia Scarisbrick, MD, Study Chair — UHB-Queen Elisabeth Medical Centre, Birmingham, United Kingdom; Emmanuella Guenova, MD, Study Chair — Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne, Switzerland
Locations (2):
- France (2):
  - CHU de Bordeaux - Groupe Hospitalier Saint-Andre - Hopital Saint-Andre, Bordeaux
  - Assistance Publique Hopitaux Paris- APHP - APHP Nord - Univ De Paris Cite - Hop. Saint Louis, Paris